CLINICAL TRIAL: NCT03682172
Title: Effect of Glucagon-like Peptide 2 on Postprandial Gallbladder Motility in Healthy Subjects
Brief Title: Effect of Glucagon-like Peptide 2 on Gallbladder Motility After a Meal in Young, Healthy Male Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-17037571
Record Dates: First submitted 2018-07-16; First posted 2018-09-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2020-06

CONDITIONS: Effect of Glucagon-like Peptide 2 on Gallbladder Motility
Keywords: Gallbladder Motility; Gallbladder Emptying; Glucagon-Like Peptide 2

STUDY DESIGN:
Intervention Model Description: It is a blinded, randomized, placebo controlled study where 15 participants receive three different 4 hour intravenous infusions of either saline (placebo), low GLP-2 (at a rate of 1pmol/kg/min) or high GLP-2 (at a rate of 10pmol/kg/min) on three different study days.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GLP-2 (10pmol/kg/min) (Experimental): A single four hour intravenous infusion with glucagon-like peptide 2 at a rate of 10pmol/kg/min
  Interventions: Drug: GLP-2 (10pmol/kg/min)
- GLP-2 (1pmol/kg/min) (Experimental): A single four hour intravenous infusion with glucagon-like peptide 2 at a rate of 1pmol/kg/min
  Interventions: Drug: GLP-2 (1pmol/kg/min)
- Placebo (Experimental): A single four hour intravenous infusion with saline water (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-2 (1pmol/kg/min) — Four hour intravenous infusion with glucagon-like peptide 2 at a rate of 1pmol/kg/min
  Arms: GLP-2 (1pmol/kg/min)
Drug: GLP-2 (10pmol/kg/min) — Four hour intravenous infusion with glucagon-like peptide 2 at a rate of 10 pmol/kg/min
  Arms: GLP-2 (10pmol/kg/min)
Drug: Placebo — Four hour intravenous infusion with saline water
  Arms: Placebo

SUMMARY:
The study will investigate the effect of the incretin hormone glucagon-like peptide 2 (GLP-2) on postprandial gallbladder motility in young, healthy, male subjects.

The study is double-blinded, randomized and placebo controlled. 15 subjects will be included. On three separate study days (A, B, C) the subjects will receive an four hour intravenous infusion with either saline (placebo), GLP-2 at a rate of 1 pmol/kg/min or GLP-2 at a rate of 10 pmol/kg/min 30 minutes after the infusion start the subject will receive a liquid meal which will stimulate gallbladder contraction.

The gallbladder volume will be determined by frequent ultrasonic scans, and blood samples will be drawn on fixed times through out the study day.

DETAILED DESCRIPTION:
Study design The primary endpoint is the incremental Area Under the Curve (iAUC) of the gallbladder Ejection Fraction % (EF) at time 0-210 minutes. Gallbladder volume will be measured during a four hour intravenous GLP-2 infusion at two different concentrations (1 pmol/kg body weight/min and 10pmol/kg body weight/min), respectively, compared to placebo after ingestion of a liquid meal in healthy, young, male subjects. The gallbladder volume will be quantified by multiple ultrasonography scans at fixed times during the experimental study days.

Gallbladder ejection fraction (EF%) will be calculated as following:

Gallbladder EF = (gallbladder volume, baseline - gallbladder volume, at a given time t) / gallbladder volume, baseline * 100. The gallbladder volume is determined by bedside ultrasonography.

15 healthy male subjects will be included according to the inclusion and exclusion criteria listed below.

Inclusion criteria:

Sex: Male Ethnicity: Caucasian Age: 18-35 years BMI: 18.5-24.9 Fasting plasma glucose: 6 mmol/l or below Glycated haemoglobin (HbA1c): 42 mmol/mol or below Haemoglobin: 8.3-10.5 mmol/l

Exclusion criteria:

First-degree relatives with type 1 or type 2 diabetes Nephropathy (serum creatinin > 130 micromole/l) Liver disease Active or recent malignant disease

A subject will participate in three study days (day A, B and C) with a minimum of 48 hours between each day. The three days will differ in regards to the intravenous infusion:

Study day A (placebo):

Subjects arrive at the laboratory after an overnight fast (10h). Two cannulas will then be inserted in the cubital veins (one in each arm) for collection of blood samples and administration of saline (placebo), respectively. The forearm from which blood samples are drawn will be wrapped in a heating pad throughout the experiment. The participant must rest 30 minutes before start of the experimental procedures.

At time -30 min, saline infusion (placebo) will be started.

At time 0 min the participant will ingest a mixed liquid meal (200 ml, 1260 kJ) mixed with paracetamol (1,500 mg) dissolved in 100 ml of water.

At time -60, -30, -15, 0, 10, 30, 50, 70, 90, 120, 150, 180 and 210 min gallbladder height, width and length will be determined by ultrasound (LOGIQ E9, GE Healthcare, Waukesha, WI, USA) for evaluation of gallbladder volume (calculated by the ellipsoid method).

Blood samples will be collected at time -45, -40, -35, -20, -5, 20, 40, 60, 80, 100, 140 and 200 min for the analysis of plasma/serum concentrations of glucose, GLP-1, GLP-2, GIP, glucagon, OXM, PYY, ghrelin, gastrin, CCK, FGF-19, insulin, C-peptide, bile acids, free fatty acids, paracetamol and triglycerides.

Experimental Day B (GLP-2 (1 pmol/kg/min)) As experimental Day A, but with infusion of GLP-2 (1 pmol/kg/min) instead of the saline infusion.

Experimental Day C (GLP-2 (10 pmol/kg/min)) As experimental Day A, but with infusion of GLP-2 (10 pmol/kg/min) instead of the saline infusion.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Male
* Age: 18-35 years
* BMI: 18,5-24,9
* Fasting plasma glucose ≤ 6 mmol/l
* Glycated haemoglobin (HbA1c) ≤ 42 mmol/mol
* Normal haemoglobin (8,3-10,5 mmol/l)
* Informed and written consent

Exclusion Criteria:

* First-degree relatives with type 1 or type 2 diabetes
* Nephropathy (se-creatinin > 130 μM and/or albuminuria)
* Liver disease (alanintransaminase (ALAT) or aspartattransaminase (ASAT) > 2 × upper normal limit)
* Active or recent malignant disease
* Treatment with medicine that cannot be paused for 1 week
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Gallbladder ejection fraction (EF%) | 0-210 minutes
  Incremental Area Under the Curve (iAUC) for gallbladder ejection fraction (EF%) at time 0-210 minutes.

SECONDARY OUTCOMES:
Glucagon | -30-200 minutes
  Incremental Area Under the Curve (iAUC) (-30;200min) of glucagon plasma concentration.
Gastric emptying | 0-200 minutes
  Gastric emptying will be determined by the by paracetamol curve following ingestion of the meal (mixed with 1500 mg paracetamol).
Time to maximum gallbladder EF% | 0-210 minutes
  Time to reach maximum gallbladder ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, phd, Principal Investigator — Clinical Metabolic Physiology, Steno Diabetes Center Copenhagen
Locations (1):
- Clinical Metabolic Physiology, Steno Diabetes Center Copenhagen, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No